CLINICAL TRIAL: NCT00284687
Title: Phase III Study Evaluating the Safety and Efficacy of Artesunate in Preemptive Treatment of Human Cytomegalovirus Disease in Stem Cell Transplant Recipients
Brief Title: Artesunate in Preemptive Treatment of Human Cytomegalovirus (CMV) in Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Institut für Klinische und Molekulare Virologie (Unknown); University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Michael Shapira, MD, Hadassah University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYS-02-HMO-CTIL
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2009-08

CONDITIONS: Cytomegalovirus Infections
Keywords: bone marrow transplantation; CMV disease
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Artesunate

INTERVENTIONS:
Drug: Artesunate — PO Artesunate

SUMMARY:
Human cytomegalovirus (HCMV) has remained a major cause of morbidity and mortality following allogeneic bone marrow or peripheral blood stem cell transplantation (SCT). The most reliable virological predictive marker for disease development is the presence of HCMV viremia. It has been further recognized that viral load, and viral load kinetics are important determinants of pathogenesis. Prior to the preventive use of antiviral agents, CMV disease occurred in 15-45% of at-risk patients and carried a high mortality rate. In the last decade, major advances in the prevention of CMV disease have occurred with the application of pp65 antigenemia and qualitative/quantitative polymerase chain reaction (PCR) assays for the rapid and sensitive diagnosis of HCMV infection, combined with preemptive antiviral treatment targeted to patients with viremia. The prevalence of early CMV disease has declined to 3% to 6% with intense antiviral drug use. All antiviral drugs currently used for the treatment of systemic HCMV infection, including ganciclovir, foscarnet, and cidofovir, target the HCMV DNA polymerase. Ganciclovir is the most widely used drug for preemptive treatment. However, ganciclovir treatment is often complicated by bone marrow toxicity with the occasional development of potentially life-threatening thrombocytopenia, granulocytopenia, and graft failure, associated with secondary bacterial and fungal infection. Another limitation of preemptive ganciclovir therapy is the requirement for intravenous administration. The currently available oral valganciclovir is not yet approved for preemptive therapy in SCT recipients, and is associated with high treatment cost. Additionally, prolonged or repeated ganciclovir treatment may lead to the development of drug resistance. The use of foscarnet and cidofovir is limited by considerable nephrotoxicity, low oral bioavailability, and high cost. Thus, there is an increasing need for new effective non-toxic, low-cost anti-HCMV drugs with high oral bioavailability.

Recently, the anti-malaria drug artesunate, which is widely used in the treatment of severe malaria, has been shown to be a highly effective inhibitor of HCMV in vitro. Artesunate exhibited similar antiviral activity (same micromolar range) to that of ganciclovir, while demonstrating no cytotoxicity. Importantly, its antiviral activity has been further demonstrated in vivo in a rat CMV model. No significant side effects were demonstrated in a number of pre-clinical and clinical studies, and artemisinin and its derivatives have been shown to be well-tolerated and safe in adults and children. Several million people have taken artemisinins to date, with no significant adverse or treatment-limiting effects being reported. Although neurotoxicity has been reported with supraphysiological doses in animals, it has not been documented in humans. Meta-analyses of malaria patients treated with artemisinins demonstrated that this drug class is safe. In rare cases, however, slight changes to haematology values have been seen, including a reduction in the number of reticulocytes as well as a slight increase in transaminase levels. These signs, however, do not generally give rise to any noticeable clinical manifestations. In rare cases, a slight but transient reduction in sinus heart rate has been observed. Abdominal cramps and mild diarrhoea have been reported at elevated doses.

Thus, one might expect a similarly high degree of safety for the potential use of artesunate as an antiviral drug for HCMV infection. Thus, oral therapy with artesunate could be a beneficial option to the current therapies for the preemptive treatment of HCMV disease in SCT recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years.
* Patients undergoing matched hematopoietic stem cell transplantation (HSCT), with antigenemia ≥ 1 positive cells/200,000 WBC, and/or CMV DNA load between 2000-10,000 copies/ml.
* Had a tri-lineage hematopoietic engraftment.
* Can take oral medications.

Exclusion Criteria:

* Not fulfilling the inclusion criteria.
* History of, or active HCMV disease*.
* Anti-CMV therapy within the past 15 days.
* Haploidentical HSCT.
* Uncontrolled graft-versus-host disease (GVHD).
* Uncontrolled or untreated bacterial, fungal, or viral (non-CMV) infection.
* Patients receiving > 2mg/kg/day prednisone treatment.
* Severe, uncontrolled diarrhea.
* Evidence of malabsorption.
* Inability to comply with study requirements.
* Known hypersensitivity to artesunate.
* Patients with relative contraindications to artesunate: preexisting cardiac or central nervous system disease
* Pregnant or lactating patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety | 60d
Efficacy | 60d

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization; Dana G Wolf, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel